CLINICAL TRIAL: NCT03334292
Title: Natural History of Wilson Disease: Registry for Patients With Wilson Disease
Brief Title: Natural History of Wilson Disease
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Wilson Disease Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1609018429
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Wilson Disease
Keywords: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Data will be collected prospectively from standard of care assessments as well as study specific assessments and entered into a central database. Some retrospective data in regards to the treatment for Wilson Disease prior to enrollment will be collected as well, if available from the medical record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the registry/repository is to provide a mechanism to store data and specimens to support the conduct of future research about Wilson disease (WD). The overall aim is to determine the optimal testing for diagnosis and parameters for monitoring treatment of WD that will aid product utilization and development.

DETAILED DESCRIPTION:
There are three aims outlined as part of this research study.

Aim 1 is to study the natural history of a carefully characterized cohort of patients with WD followed longitudinally at Centers of Excellence for WD in the United States and in the United Kingdom.

Aim 2 seeks to evaluate parameters for diagnosis and treatment monitoring for patients on chelation therapy and zinc treatment for their WD. Data gathered in Specific aim 1 will be used for analyzing the components of the diagnostic scores for patients.

Aim 3 is intended to determine whether a composite index or a biomarker can be used as surrogate marker for treatment monitoring for current patients on therapy that can be used for future patient treatment trials.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of WD
* Able and willing to provide informed consent for adults (Parental/guardian permission (informed consent) and if appropriate, child assent for participants <18 (or per local Institutional Review Board (IRB) regulation)

Exclusion Criteria:

* Diagnosis of WD has been excluded
* Unwilling to provide informed consent or assent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients being evaluated for or with a diagnosis of WD who are willing to participate in the registry at designated study sites around the United States and in the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Create registry for Wilson disease | 5 Years
  This outcome is a binary 'yes/no' outcome as to whether or not this study can successfully create a repository with the intent to store data and specimens to support the conduct of future research on Wilson disease.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Advent Health, Orlando, Florida
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- Royal Surrey Country Hospital, Guildford, Surrey, United Kingdom